CLINICAL TRIAL: NCT04236752
Title: Stereotactic Pelvic Brachytherapy With HDR Boost for Dose Escalation in High Tier Intermediate and High Risk Prostate Cancer (SPARE)
Brief Title: Stereotactic Pelvic Brachytherapy With HDR Boost for Dose Escalation in High Tier Intermediate and High Risk Prostate ca
Acronym: SPARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Prostate Cancer Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPARE
Record Dates: First submitted 2019-05-31; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: HIGH RISK PROSTATE CANCER

STUDY DESIGN:
Intervention Model Description: HDR Brachytherapy Boost of 15Gy to the prostate followed by Stereotactic Ablative Body Radiation (SBRT) 25 Gy in 5 fractions, once weekly to prostate, SVs and pelvic lymph nodes + 6-18 months of ADT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm radiotherapy (Experimental): HDR Brachytherapy Boost of 15Gy to the prostate followed by Stereotactic Ablative Body Radiation (SBRT) 25 Gy in 5 fractions, once weekly to prostate, SVs and pelvic lymph nodes + 6-18 months of ADT
  Interventions: Radiation: Stereotactic Ablative Body Radiation (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiation (SBRT)

SUMMARY:
HDR brachytherapy in conjunction with pelvic SABR in high tier intermediate and high risk prostate cancer patients can provide a safe and effective means of radiotherapy dose escalation.

Utilizing multiparametric MRI to focally boost the dominant intraprostatic lesion during HDR brachytherapy is safe and feasible.

DETAILED DESCRIPTION:
HDR brachytherapy:

Under general anesthetic, prostate will be implanted transperineally using up to 18 catheters. Three gold seed fudicials will also be implanted transperineally at base, midgland and apex forSABR treatment. Prostate will be contoured as Clinical Target Volume (CTV) on the transrectal ultrasound (TRUS) based ONCENTRA planning system. Rectum and urethra will be contoured as organs at risk. 15Gy will be prescribed to CTV as the MPD (minimal Peripheral Dose).

Treatment Delivery-SABR There will be a 2 week interval between HDR and SABR component to allow for normal tissue recovery and radiotherapy planning time. Daily image guidance will be performed using the implanted fiducials to calculate patient shifts to ensure proper positioning. Post-treatment images will be taken to estimate intrafraction motion.

Androgen Deprivation Therapy Twelve to 18 months of luteinizing-hormone releasing hormone agonists (LHRHa) will be used. Anti-androgen and neoadjuvant LHRHa can be used according to physician discretion

Follow-Up and Toxicity Assessment Time zero will be the start of radiotherapy. Baseline rectal and urinary function will be recorded using common toxicity criteria adverse effect (CTCAE v3.0) and Expanded prostate Cancer Index Composite (EPIC). CTCAE v3.0 and EPIC assessments will be done at weeks 3, 5 and 12 weeks. Bloodwork (PSA and testosterone), quality of life (EPIC) and late GI and GU toxicity evaluation (using the RTOG/EORTC Late Radiation Morbidity Scheme) will be performed every 6 months for the first 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Men >18 years
* Histologically confirmed prostate adenocarcinoma (centrally reviewed)
* High tier intermediate risk defined as :

Clinical stage T1-T2c AND PSA 10-20ng/ml AND {PSA>10ng/ml AND (T2b-2c Or Gleason 7)} OR Gleason 4+3

-High-risk prostate cancer, defined as at least one of: Clinical stage T3, OR Gl 8-10, OR PSA > 20 ng/mL

Inclusion Criteria:

* Prior pelvic radiotherapy
* Anticoagulation medication (if unsafe to discontinue for gold seed insertion)
* Diagnosis of bleeding diathesis
* Large prostate (>50cm3) on imaging
* No evidence of castrate resistance (defined as PSA < 3 ng/ml while testosterone is < 0.7 nmol/l. Patients could have been on combined androgen blockade but are excluded if this was started due to PSA progression.
* Definitive regional or distant metastatic disease on staging investigations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute GI and GU toxicities | Baseline (start of treatment) to 6 weeks post completion of Radiation treatment
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v3.0, Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks. This will be calculated using the F distribution method (exact confidence limits).

SECONDARY OUTCOMES:
Late GI and GU RTOG toxicities | 6 months post start of treatment to end of 5 year follow up post completion of treatment
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v3.0, Change From 6 months post treatment to end of 5 year follow up. This will be calculated using the F distribution method (exact confidence limits).
Quality of Life outcome- EPIC | Baseline ( start of treatment) to end of 5 year follow up post completion of treatment
  Quality of life using the Expanded Prostate Cancer Index Composite (EPIC) questionnaire.
Biochemical disease-free survival | Baseline ( start of treatment) to end of 5 year follow up post completion of treatment
  Biochemical disease-free survival post treatment
Quality of Life outcome- EQ5D | Baseline to end of 5 year follow up post completion of treatment
  Assess the impact of modifiable life style factors on radiation toxicity as well as Determine the health preference values using the EQ5D(EQ-5D is the name of the instrument and is not an acronym.)

OTHER OUTCOMES:
Quality of Life outcome- PORPUS-U | Baseline ( start of treatment) to end of 5 year follow up post completion of treatment
  Assess the impact of modifiable life style factors on radiation toxicity as well as Determine the health preference values using the PORPUS -U(PORPUS-U is the name of the instrument and is not an acronym.)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontairo, Canada

IPD SHARING:
Plan to Share IPD: No
Overall study data will be available thru publications. Individual Participants Data will not be made public.